CLINICAL TRIAL: NCT04854031
Title: Stream Segregation and Speech Recognition in Noise in Individuals With Cochlear Implants
Status: Completed | Type: Observational
Sponsor: Father Flanagan's Boys' Home (Other)
Responsible Party: Principal Investigator, Adam Bosen, Director, Auditory Perceptual Encoding Laboratory, Father Flanagan's Boys' Home
Other Study IDs: 5P20GM109023-07 (NIH)
Record Dates: First submitted 2021-04-16; First posted 2021-04-22 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Cochlear Implants
MeSH Terms: interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Cochlear Implant Recipients: 30 participants who lost their hearing and received one or two cochlear implants as adults will participate in this study. We will include unilaterally and bilaterally implanted individuals listening with their everyday hearing configuration. Individuals with residual acoustic hearing better than 60 A-weighted decibels at any audiometric frequency will be excluded. Participants will range in age between 19 and 80 years old, although most are expected to be within 50 - 75 years of age.
  Interventions: Device: Cochlear Implants

INTERVENTIONS:
Device: Cochlear Implants — Individuals with cochlear implants will be tested on their hearing ability. Auditory recordings of speech will be played to participants from a loudspeaker. Recordings will be edited to add competing noise sources and to adjust talker voice pitch. Synthetic sounds will be manipulated to control auditory cue salience in detection tasks.

SUMMARY:
Individuals with cochlear implants will complete tasks which measure auditory resolution, working memory, stream segregation, and speech recognition in the presence of competing speech using their everyday clinical device settings. The relationship between these tasks will be examined to identify the factors which predict successful speech recognition in the presence of competing speech.

DETAILED DESCRIPTION:
Individuals with cochlear implants struggle to understand speech in the presence of competing talkers because they have trouble segregating auditory streams. The premise of this project is that individual differences in auditory resolution and cognitive ability across individuals with cochlear implants determine the extent to which they can segregate auditory streams from one another and hear out target speech embedded in competing talkers. Our goal is to test whether the link between speech recognition in noise and individual differences in auditory resolution and working memory in individuals with cochlear implants is due to the limitations that these individual differences place on stream segregation. The outcome measure to be predicted is sentence recognition in two-talker babble. Previous work has found that spectral and temporal modulation detection thresholds (measures of auditory resolution) and performance on the reading span task (a measure of working memory that is closely linked to fluid intelligence) are predictors of speech recognition in quiet. To account for these sources of variability in speech recognition, we will verify that these tasks jointly predict individual differences in sentence recognition in quiet. Adding competing talkers during the speech recognition task will introduce additional variability beyond the variability of speech recognition in quiet. We hypothesize that this additional variability with competing talkers should be predicted by individual differences in stream segregation ability, which will in turn be predicted by auditory resolution and working memory. Obligatory and voluntary stream segregation ability will be measured using rapidly presented digit sequences manipulated to have alternating fundamental frequencies (F0) for each digit. Participants will resist integration and repeat back only the digits presented with the higher F0. The magnitude of the F0 alternation will be manipulated to control the difficulty of segregating streams. The predicted relationship between stream segregation and sentence recognition will be tested for auditory resolution and working memory in independent and combined models. Completing this goal will identify the auditory and cognitive factors that support stream segregation in post-lingually deafened adults with cochlear implants. This identification will enable development of cochlear implant design and rehabilitation strategies to facilitate stream segregation in these patients as well as investigation of the developmental trajectories of these factors in children with cochlear implants. We plan to implement this study in at-home testing conditions to avoid risking coronavirus disease 2019 transmission in the lab, so this work will also determine the feasibility of at-home testing of individuals with cochlear implants. At-home testing would expand the amount and diversity of participants we are able to recruit for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Has at least one cochlear implant.
* Lost their hearing during adulthood.
* Native English speaker.

Exclusion Criteria:

* Cognitive impairment

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Cochlear Implants who are enrolled in the Boys Town National Research Hospital research database
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam K Bosen, Principal Investigator — Father Flanagan's Boys' Home
Locations (1):
- Boys Town National Research Hospital, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified results from all experimental tasks will be made publicly available through the Open Science Framework. Relevant demographic information will be provided for each participant.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Following completion of the study and publication of results in a peer-reviewed journal.
Access Criteria: Publicly available

RESULTS

PARTICIPANT FLOW:
Groups:
- Cochlear Implant Recipients: 8 participants who lost their hearing and received one or two cochlear implants as adults will participate in this study. We will include unilaterally and bilaterally implanted individuals listening with their everyday hearing configuration. Individuals with residual acoustic hearing better than 60 A-weighted decibels at any audiometric frequency will be excluded. Participants will range in age between 19 and 80 years old, although most are expected to be within 50 - 75 years of age.
  Cochlear Implants: Individuals with cochlear implants will be tested on their hearing ability. Auditory recordings of speech will be played to participants from a loudspeaker. Recordings will be edited to add competing noise sources and to adjust talker voice pitch. Synthetic sounds will be manipulated to control auditory cue salience in detection tasks.
Period: Overall Study
Arm/Group | Cochlear Implant Recipients
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 67 [57 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Speech Recognition
Description: The metric for speech recognition is the percentage of Perceptually Robust English Sentence Test Open-set (PRESTO) sentence keywords that were correctly repeated in order.
Time Frame: Up to 30 minutes in each of two listening conditions.
Population: The entire population
Measure: Mean (Full Range); unit: percentage of keywords correct
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 8
percentage of keywords correct
  In quiet | 62 [30 to 80]
  In +10 decibel target-to-masker ratio two-talker babble | 22 [9 to 28]

2. Primary Outcome: Temporal Modulation Detection Threshold
Description: The metric for temporal modulation detection is the modulation depth relative to 100% modulation which the participant can detect 71% of the time.
Time Frame: Up to 30 minutes
Population: The entire population
Measure: Mean (Full Range); unit: decibels relative to 100% modulation
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 8
decibels relative to 100% modulation | -3.1 [-6.2 to -0.4]

3. Primary Outcome: Spectral Modulation Detection Thresholds
Description: The metric for spectral modulation detection is the magnitude of the peak-to-valley ratio of the spectrally modulated stimulus which the participant can detect 71% of the time.
Time Frame: Up to 30 minutes
Population: The entire population
Measure: Mean (Full Range); unit: decibels peak-to-valley ratio
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 8
decibels peak-to-valley ratio | 12.8 [4.8 to 34]

4. Primary Outcome: Reading Span Task Performance
Description: The outcome is the percentage of letters recalled in the correct position across all trials, out of a total of 75 letters.
Time Frame: Up to 20 minutes
Population: The entire population
Measure: Mean (Full Range); unit: Percentage of Letters Recalled
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 8
Percentage of Letters Recalled | 57 [33 to 91]

5. Primary Outcome: Digit Span Task Performance
Description: The outcome is the total percentage of digits recalled in the correct position across all trials, out of a maximum of 220.
Time Frame: Up to 20 minutes
Population: The entire population
Measure: Mean (Full Range); unit: percentage of digits recalled
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 8
percentage of digits recalled | 64 [49 to 92]

6. Primary Outcome: Free Recall Task Performance
Description: The outcome is the average number of words recalled from each list, with a possible maximum of 12.
Time Frame: Up to 10 minutes
Population: The entire population
Measure: Mean (Full Range); unit: average number of words recalled
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 8
average number of words recalled | 3.3 [2.1 to 4.8]

7. Primary Outcome: Digit Updating Task Performance
Description: The outcome is the percentage of numbers correctly recalled across boxes, out of a total of 49.
Time Frame: Up to 20 minutes
Population: The entire population
Measure: Mean (Full Range); unit: Percentage of numbers recalled
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 8
Percentage of numbers recalled | 57 [18 to 86]

8. Primary Outcome: Running Digit Span Task Performance
Description: The outcome is the average number of digits recalled in the correct position relative to the last item in the sequence across lists.
Time Frame: Up to 15 minutes
Population: The entire population
Measure: Mean (Full Range); unit: Average number of digits recalled
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 8
Average number of digits recalled | 2.4 [1.1 to 3.9]

9. Primary Outcome: Stream Segregation
Description: The metric for stream segregation is the percent change in digit recall that occurs when voice pitch differs from the distractor digits (85, 120, and 150 Hz) relative to when voice pitch between target and distractor digits is the same (200 Hz).
Time Frame: Up to 1 hour
Population: The entire population
Measure: Mean (Full Range); unit: Percentage difference in digits recalled
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 8
Percentage difference in digits recalled
  85 Hz Target, 200 Hz Distractor | 12.5 [-20 to 43]
  120 Hz Target, 200 Hz Distractor | 12.5 [-35 to 43]
  150 Hz Target, 200 Hz Distractor | 16 [-8 to 42]

ADVERSE EVENTS:
Time Frame: Through study completion, a maximum of 5 hours per participant.
Arm/Group | Cochlear Implant Recipients
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Recruiting difficulties lead to a smaller total number of participants than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT04854031/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT04854031/SAP_001.pdf